CLINICAL TRIAL: NCT00294567
Title: Azelnidipine and Amlodipine Anti-Coronary Atherosclerotic Trial in Hypertensive Patients Undergoing Coronary Intervention by Serial Volumetric Intravascular Ultrasound Analysis in Junten Medical University (ALPS-J)
Brief Title: Azelnidipine Anti-Coronary Atherosclerotic Trial in Hypertensive Patients by Serial Volumetric IVUS Analysis(ALPS-J)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juntendo University (Other)
Collaborators: Japan Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHF-17NOV2005
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2008-10

CONDITIONS: Hypertension; Coronary Atherosclerosis
Keywords: Hypertension; PCI; Calcium Channel Blockers; IVUS; Plaque
MeSH Terms: conditions — Hypertension; Coronary Artery Disease; Plaque, Amyloid | interventions — Calcium Channel Blockers; Amlodipine; azelnidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Amlodipine
  Interventions: Drug: Calcium channel blockers (amlodipine, azelnidipine)
- 2 (Active Comparator): Azelnidipine
  Interventions: Drug: Calcium channel blockers (amlodipine, azelnidipine)

INTERVENTIONS:
Drug: Calcium channel blockers (amlodipine, azelnidipine) — Drug: amlodipine Drug: azelnidipine

SUMMARY:
In patients with hypertension who undergo elective PCI, the effects of long-term administration of Calblock (azelnidipine) on plaque volume will be determined quantitatively by 3D-IVUS and compared with those of amlodipine besilate (Norvasc or Amlodin).

DETAILED DESCRIPTION:
Clinical studies have demonstrated that calcium antagonists can reduce cardiovascular events in patients with coronary artery disease. Recently, suppression of the development of coronary atherosclerotic plaque by calcium antagonists has been reported as one of the mechanisms involved. Thus, calcium antagonists have been promising strategy for preventing the progression of the coronary atherosclerosis. Various calcium antagonists are clinically available at present and these drugs may differ from each other with respect to the anti-atherosclerotic effects. Consequently, we plan to perform the ALPS-J study to compare the effects of two long-acting calcium antagonists, azelnidipine and amlodipine, on plaque quantitatively by IVUS. In this study, azelnidipine (16 mg/day) or amlodipine besilate (5 mg/day) will be administered to patients with hypertension for 48 weeks after elective PCI. The plaque volume will be measured in each patient by IVUS at the time of PCI and 48 weeks after PCI. Percent change in plaque volume from the baseline value will be used as the primary endpoints for evaluation of efficacy. We plan to enroll 100 patients in each group for a total of 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 and 79 years (at the time of giving informed consent).
* Sex: Either sex.
* Admission status: Outpatients.
* Patients requiring treatment for hypertension according to the JSH 2004 hypertension therapy guidelines before beginning this study
* Patients who have not used any calcium antagonists for at least 4 weeks before the beginning of this study.
* Patients who are scheduled to undergo elective PCI.

Exclusion Criteria:

* Patients with acute coronary syndrome (ACS).
* Patients who have experienced Q-wave myocardial infarction within 4 weeks before beginning this study.
* Patients with renal dysfunction (serum creatinine >2.0 mg/dL).
* Patients in whom PCI is unsuccessful.
* Patients with cardiogenic shock.
* Patients with moderate or severe congestive heart failure.
* Patients with 50% or more stenosis of the main trunk of the left coronary artery.
* Patients with other problems whom the investigator considers unsuitable for this study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percent change in plaque volume from the baseline value. (IVUS) Percent change in plaque volume = (plaque volume after 48 weeks of drug administration - baseline plaque volume) / baseline plaque volume | 48Weeks

SECONDARY OUTCOMES:
Change of plaque volume from the baseline value. (IVUS) Amount change and percent change in Minimal lumen diameter and % stenosis. (Quantitative Coronary Analysis) Change of intimal thickening volume in-stent. | 48Weeks
Correlativity of plaque volume and inflammatory laboratory parameters (hs-CRP, MCP-1, PTX-3) Correlativity of laboratory parameters and blood pressure. Correlativity of plaque volume and antioxidant laboratory parameters (LPO, 8-isoprostane) | 48Weeks
The following treatments and incidence of events, Changes from baseline of laboratory parameters (TC, LDL-C,TG, HDL-C, hs-CRP, MCP-1, LPO, 8-isoprostane, PTX-3) after 48 weeks of drug administration. Correlativity of plaque volume and blood pressure. | 48Weeks

CONTACTS AND LOCATIONS:
Overall Officials: HIROYUKI MD DAIDA, Study Chair — Director of Cardiology Professor of Medicine
Locations (1):
- Department of Cardiology, Juntendo University School of Medicine, Tokyo, Japan

REFERENCES:
- [Derived] Miyauchi K, Daida H. [Azelnidipine and amlodipine anti-coronary atherosclerosis trial in hypertensive patients undergoing coronary intervention by serial volumetric intravascular ultrasound analysis in Juntendo Medical University]. Nihon Naika Gakkai Zasshi. 2012 Oct 10;101(10):3002-11. doi: 10.2169/naika.101.3002. No abstract available. Japanese. PMID 23214115
- [Derived] Kojima T, Miyauchi K, Yokoyama T, Yokoyama K, Kurata T, Suwa S, Kawamura M, Tamura H, Okazaki S, Inoue K, Fujiwara Y, Sumiyoshi M, Tanimoto K, Nakazato Y, Yamagami S, Hiro T, Komiyama N, Daida H. Azelnidipine and amlodipine anti-coronary atherosclerosis trial in hypertensive patients undergoing coronary intervention by serial volumetric intravascular ultrasound analysis in Juntendo University (ALPS-J). Circ J. 2011;75(5):1071-9. doi: 10.1253/circj.cj-11-0141. Epub 2011 Apr 7. PMID 21471671